CLINICAL TRIAL: NCT04316806
Title: Efficacy of a Probiotic Formula in Reducing Small Intestinal Bacterial Overgrowth (SIBO) in Patients With Irritable Bowel Syndrome (IBS)
Brief Title: Effect of a Probiotic Formula on Reducing SIBO in IBS Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator changed his job
Sponsor: AB Biotics, SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Probiotic_IBS+SIBO
Record Dates: First submitted 2020-03-03; First posted 2020-03-20 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-02

CONDITIONS: Irritable Bowel Syndrome; Small Intestinal Bacterial Overgrowth
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Probiotics; Rifaximin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Treatment with probiotic formula
  Interventions: Dietary Supplement: Probiotic
- Antibiotic (Other): Treatment with antibiotic rifaximin
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic (dietary supplement) administrated once daily (u.i.d) for 8 weeks (3 billion cfus per day)
  Arms: Probiotic
Drug: Rifaximin — Antibiotic rifaximin consisting 400 mg capsules administrated twice daily (b.i.d) for 1week.
  Arms: Antibiotic

SUMMARY:
This randomized study evaluates the effectiveness of the a probiotic formula, compared with the antibiotic rifaximin, in the treatment of Small Intestinal Bacterial Overgrowth (SIBO) in Irritable Bowel Syndrome (IBS) patients.

DETAILED DESCRIPTION:
Irritable Bowel Syndrome (IBS) is a functional gastrointestinal disease in which recurrent abdominal pain is associated with defecation or a change in bowel habits. Disordered bowel habits are typically present (ie, constipation, diarrhea, or a mix of constipation and diarrhea), as are symptoms of abdominal bloating/distention.

IBS pathophysiology is multifactorial and may include alterations of the gut microbiota, food intolerances and Small Intestinal Bacterial Overgrowth (SIBO). However, SIBO is a distinct entity than IBS, as patients can present SIBO without IBS. SIBO is diagnosed based on objective tests (breath test or microbial culture of duodenal aspirate) while IBS is a functional syndrome, diagnosed on symptoms (Rome-IV criteria).

A probiotic formula composed of strains Pediococcus acidilactici CECT 7483 and Lactobacillus plantarum CECT 7484 and CECT 7485 was previously shown to improve quality of life in patients with IBS.

Rifaximin is a a non-absorbable antibiotic commonly used for the treatment of SIBO.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with IBS according to Rome IV criteria (Lacy et al. Gastroenterology 2016) and with SIBO according to North American Consensus (Rezaie et al., Am J Gastroenterol. 2017), providing Informed Consent.

Patients taking set doses of Proton Pump Inhibitors (PPIs) or antispasmodics can be included.

Exclusion Criteria:

* Use of antibiotics in the 4 weeks before study initiation.
* Use of probiotics in the 2 weeks before study initiation.
* Use of loperamide or other prokinetics in the week before study initiation.
* Use of Plantago ovata, lactulose or other laxans in the week before study initiation.
* Use of antidepressants.
* Suspicion or confirmed diagnose of coeliac disease, inflammatory bowel disease (IBD), symptomatic diverticulosis/diverticulitis, or endometriosis.
* Previous intestinal surgery, except appendectomy and herniorrhaphy.
* Short bowel syndrome or pancreatitis.
* Concomitant treatment with immunosuppressors, oncologic disease, severe cardiovascular disease, positive for HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV).
* Other conditions that can interfere with the effect of probiotic.
* Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
SIBO | 0 and 4 weeks
  SIBO evolution determined by changes in exhaled H2 and methane (CH4) levels after ingestion of lactulose (25 g)

SECONDARY OUTCOMES:
Gut microbiota | 0 and 4 weeks
  Intestinal microbiota composition studied by metagenomics analysis from faecal samples
IBS severity | 0, 4 and 8 weeks
  Measurement of IBS severity by Irritable Bowel Syndrome-Severity Score (IBSSS), ranging from 0 to 500 (<75, remission; 75-175, mild; 175-300, moderate; >300, severe cases)
Intestinal related anxiety | 0, 4 and 8 weeks
  Measurement of gastrointestinal specific anxiety by Visceral Sensitivity Index (VSI), 15 questions rated from 1 to 6. Higher ratings represent greater severity (min score= 15, max score= 90).
Global improvement after treatment | 8 weeks
  Measured with on one question with 7 possible answers: (1) much worse, (2) moderately worse, (3) slightly worse, (4) unchanged, (5) slightly better, (6) moderately better, or (7) much better.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Bofill Clinic, Girona, Spain

IPD SHARING:
Plan to Share IPD: No